CLINICAL TRIAL: NCT05994053
Title: Neuromodulation for a Novel OCD Biomarker and Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Robert Reinhart, Associate Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4555
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: OCD

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active HD-tACS (Active Comparator): HD-tACS of OFC
  Interventions: Device: high definition transcranial alternating current stimulation
- Sham HD-tACS (Sham Comparator): HD-tACS of OFC
  Interventions: Device: high definition transcranial alternating current stimulation

INTERVENTIONS:
Device: high definition transcranial alternating current stimulation — low intensity alternating current to OFC

SUMMARY:
Although multiple treatments for OCD exist, slow symptom decrease, high remission, and significant side effects for some OCD patients limit their efficacy. More research into the precise neural mechanisms and linked cognitive functions in OCD is also necessary. To address both concerns, this study by Dr. Reinhart and his team will test a new, non-invasive, and well-tolerated neuromodulation method for reducing OCD symptoms, based on reward-related rhythms of the orbitofrontal cortex (OFC; a brain region responsible for reward, decision making and other crucial functions that is affected by OCD). This proposal is based on highly encouraging preliminary data in both subsyndromal and treatment-resistant populations that shows rapid reductions in OCD behaviors that last at least 1-3 months. Using high-definition transcranial alternating current stimulation (HD-tACS) guided by EEG brain wave recordings, the study will test whether repetitive modulation of relevant rhythm activity in the OFC can lead to rapid (within five days) and sustainable (up to three months) OCD symptom reduction. This research aims to increase knowledge of OCD and development of effective treatment with minimal side effects.

ELIGIBILITY:
Inclusion Criteria:

(1) a primary DSM-5 diagnosis of OCD, (2) a score of 16 or greater on the YBOCS (3) at least 18 years of age; and (4) willingness and ability to provide informed consent and comply with the requirements of the study protocol.

Exclusion Criteria:

(1) a lifetime history of bipolar or psychotic disorders; (2) history of Tourette syndrome; (3) psychosurgery; (4) substance abuse or dependence (other than nicotine) in the past 3 months; (5) organic brain syndrome, mental retardation or other potentially interfering cognitive dysfunction; (6) severe depression (MADRS score of 30 or greater); (7) suicidal risk as determined by moderate or greater score on the Columbia Suicide Severity Rating Scale (C-SSRS); (8) pregnancy or lactation; (9) changes to pharmacotherapy for OCD or the initiation of cognitive-behavior therapy within the last 3 months; and (10) specific to the tACS and EEG procedures no metal implants in head, any implanted electronic devices, any skin sensitivity, color blindness or impaired vision despite correction, claustrophobia, and any history of epilepsy or neurological disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
YBOCS | day 5 of intervention
  There are 10 YBOCS questions scored 0 to 4. The total Y-BOCS score is the sum of items 1-10. A higher score is worse.

SECONDARY OUTCOMES:
YBOCS | 1 month after intervention
  There are 10 YBOCS questions scored 0 to 4. The total Y-BOCS score is the sum of items 1-10. A higher score is worse.
YBOCS | 2 months after intervention
  There are 10 YBOCS questions scored 0 to 4. The total Y-BOCS score is the sum of items 1-10. A higher score is worse.
YBOCS | 3 months after intervention
  There are 10 YBOCS questions scored 0 to 4. The total Y-BOCS score is the sum of items 1-10. A higher score is worse.
EEG beta-gamma rhythms | day 5 of intervention
EEG beta-gamma rhythms | 1 month after intervention
EEG beta-gamma rhythms | 2 months after intervention
EEG beta-gamma rhythms | 3 months after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University Center for Anxiety and Related Disorders (BU-CARD), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No